CLINICAL TRIAL: NCT06467695
Title: The Effect of MRI-Guided Transcranial Direct Current Stimulation on Cognitive and Affective Symptoms in Persons With Parkinson's Disease and Controls
Brief Title: Low Voltage Electrical Stimulation for Depression in Parkinson's Patients
Acronym: LVESDIPP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Alabama (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2128181
Record Dates: First submitted 2024-05-01; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Parkinson Disease; Depressive Symptoms
Keywords: Direct Transcranial Current Stimulation
MeSH Terms: conditions — Parkinson Disease; Depression

STUDY DESIGN:
Intervention Model Description: Participants (n = 40) will be either in the Parkinson's Group (n = 20) or the No Parkinson's Control (N = 20). All patients will be randomly assigned to receive either tDCS or SHAM tDCS.
Who Masked: Participant
Masking Description: Participants will not be told whether they are receiving tDCS or SHAM tDCS in order to reduce subject expectancy bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrical Stimulation (experimental) (Experimental): Transcranial Direct Current Stimulation will be administered in a high definition anodal montage at 2 milliamps with anode over T3 (adjusted for each participant) and cathode in an equidistance ring around it with 4 return electrodes. There will be 13 minutes of active stimulation followed by a twenty minute delay, followed by 13 minutes of stimulation. Participants in the pilot study will be administered 2 mA of current at a steady state with a 30 second ramp-up and ramp-down period at the beginning and end of each 13 minute stimulation interval.
  Interventions: Device: BIOPAC Stimsola
- Sham Stimulation (Sham Comparator): For the sham TDCS condition, 10 participants will receive receive sham tDCS consisting of 30 seconds of ramp-up and then the amperage will be reduced to 0 for the remainder of the session.
  Interventions: Device: BIOPAC Stimsola Sham (zero amps)

INTERVENTIONS:
Device: BIOPAC Stimsola — Transcranial Electrical Stimulator
  Arms: Electrical Stimulation (experimental)
Device: BIOPAC Stimsola Sham (zero amps) — Transcranial Electrical Stimulator set to 0 amps
  Arms: Sham Stimulation

SUMMARY:
The goal of this clinical trial is to determine the relative efficacy of fMRI model guided Transcranial Direct Current Stimulation (mgTDCS) in improving the depressive symptoms of patients with Parkinson's Disease (PD). The main questions it aims to answer are: 1) Can the use of mgTDCS significantly improve the self-reported level of depression and apathy in patients with PD from pre-intervention to post-intervention compared to a sham control? 2) Can the use of mgTDCS significantly normalize the cortical eeg alpha asymmetry so commonly seen in depressed patients compared to sham mgTDCS? 3) Can the use of mgTDCS significantly improve scores on neuropsychological tests of working memory?

DETAILED DESCRIPTION:
This study seeks to expand the growing body of literature on the use of a particular type of low voltage electrical stimulation known as Transcranial Direct Current Stimulation (TDCS) to reduce the symptoms of Parkinson's Disease (PD). One common disorder that can result from, and/or be exacerbated by PD is Major Depressive Disorder. In particular, apathy has been noted as a common and detrimental component for those with PD. While many studies have been performed on PD patients using TDCS, the consensus in the literature is that results are widely variable.

Participants will:

* complete self-report measures and neuropsychological tests
* undergo eeg recording pre and post intervention
* participate in 15, 46 minute sessions (2 13 minute stimulation sessions with 20 minutes of rest between) of mgTDCS over the course of 4-5 weeks Researchers will compare active mgTDCS to Sham mgTDCS to see if active mgTDCS is more effective. A non Parkinson's group of depressed controls who are age-matched to the PD patients will serve to determine if treatment effects are specific to PD or generalize to depression more generally.

ELIGIBILITY:
Inclusion Criteria:

* 19 to 65 years in age.
* Parkinson's Group must have a physician dx of Parkinson's Disease
* Must meet exhibit elevated levels of depression on the Beck Depression Inventory (scores of 20 or above).
* Must be willing and able to travel of the Psychology Department for EEG and tDCS sessions.
* Participants who have undergone surgery for Deep Brain Stimulation implantation may be enrolled if advised to and monitored by their physician.
* Read and understand spoken English.

Exclusion Criteria:

* No history of or being treated for epilepsy or other seizure disorders.
* No history of penetrating head wounds or TBI greater than mild TBI.
* No history of atypical Parkinson's

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-28 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory (BDI) Pre-post change score | One at Day 1 and one after 15 sessions of training, typically 4 weeks after study start.
  The BDI, a self-report measure for assessing depression, has high internal consistency (Cronbach's alpha > .90) and good test-retest reliability.
Alpha band power pre-post change score | One at Day 1 and one after 15 sessions of training, typically 4 weeks after study start.
  Alpha band power from pre-post eeg records will be assessed for power changes at frontal sites.
RBANS Working Memory | One at Day 1 and one after 15 sessions of training, typically 4 weeks after study start.
  Digit Span and Story Memory subtests will be used to determine changes in working memory.

SECONDARY OUTCOMES:
PDQ-39 | One at Day 1 and one after 15 sessions of training, typically 4 weeks after study start.
  This a common measure to assess patient quality of life in Parkinson Disease patients involved in research.

CONTACTS AND LOCATIONS:
Overall Officials: John Shelley-Tremblay, PhD, Principal Investigator — 2514606883

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Del Felice A, Castiglia L, Formaggio E, Cattelan M, Scarpa B, Manganotti P, Tenconi E, Masiero S. Personalized transcranial alternating current stimulation (tACS) and physical therapy to treat motor and cognitive symptoms in Parkinson's disease: A randomized cross-over trial. Neuroimage Clin. 2019;22:101768. doi: 10.1016/j.nicl.2019.101768. Epub 2019 Mar 18. PMID 30921609
- [Background] Brak IV, Filimonova E, Zakhariya O, Khasanov R, Stepanyan I. Transcranial Current Stimulation as a Tool of Neuromodulation of Cognitive Functions in Parkinson's Disease. Front Neurosci. 2022 Jul 12;16:781488. doi: 10.3389/fnins.2022.781488. eCollection 2022. PMID 35903808
- [Background] Broeder S, Vandendoorent B, Hermans P, Nackaerts E, Verheyden G, Meesen R, de Xivry JO, Nieuwboer A. Transcranial direct current stimulation enhances motor learning in Parkinson's disease: a randomized controlled trial. J Neurol. 2023 Jul;270(7):3442-3450. doi: 10.1007/s00415-023-11669-3. Epub 2023 Mar 23. PMID 36952012
- [Background] Broeder S, Nackaerts E, Heremans E, Vervoort G, Meesen R, Verheyden G, Nieuwboer A. Transcranial direct current stimulation in Parkinson's disease: Neurophysiological mechanisms and behavioral effects. Neurosci Biobehav Rev. 2015 Oct;57:105-17. doi: 10.1016/j.neubiorev.2015.08.010. Epub 2015 Aug 20. PMID 26297812
- [Background] de Oliveira PCA, de Araujo TAB, Machado DGDS, Rodrigues AC, Bikson M, Andrade SM, Okano AH, Simplicio H, Pegado R, Morya E. Transcranial Direct Current Stimulation on Parkinson's Disease: Systematic Review and Meta-Analysis. Front Neurol. 2022 Jan 10;12:794784. doi: 10.3389/fneur.2021.794784. eCollection 2021. PMID 35082749